CLINICAL TRIAL: NCT01332916
Title: Impact of Cancer on Memory Functioning: Understanding Disorders Using Approaches in Neuropsychology and Neuroimaging
Acronym: CANMEM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of patient
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Pr Florence JOLY-LOBBEDEZ, Centre François Baclesse
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CANMEM
Record Dates: First submitted 2011-04-08; First posted 2011-04-11 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer; Healthy
Keywords: No metastatic breast cancer; cognitive troubles; adjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients aged 45 and over group (Experimental): patients aged 45 and over with breast cancer and should receive an adjuvant chemotherapy
  Interventions: Procedure: cognitive tests and cerebral IRM
- healthy volunteers (controls) aged 45 and over (Active Comparator): healthy volunteers (controls) aged 45 and over
  Interventions: Procedure: cognitive tests and cerebral IRM

INTERVENTIONS:
Procedure: cognitive tests and cerebral IRM — cognitive tests and cerebral IRM
  Arms: patients aged 45 and over group
Procedure: cognitive tests and cerebral IRM — cognitive tests and cerebral IRM
  Arms: healthy volunteers (controls) aged 45 and over

SUMMARY:
The purpose of this study is to investigate memory problems in patients with cancer.

ELIGIBILITY:
Inclusion Criteria for patients:

* Patients aged 45 and over
* Patients from Grade 3 'end of primary schooling "minimum (scale Barbizet)
* Non-Metastatic Breast Cancer
* Adjuvant Chemotherapy: FEC, including Docetaxel Protocols
* No major cognitive impairment
* No previous neurological
* Lack of personality disorders and psychiatric disorders evolutionary
* Having signed the informed consent of study participation

Inclusion Criteria for control group:

* Women from the general population aged 45 and over, and matched in age and cultural level in patients
* Topics of Grade 3 'end of primary schooling "minimum (scale Barbizet)
* No prior cancer
* No major cognitive impairment
* No previous neurological
* Lack of personality disorders and psychiatric disorders evolutionary
* Participating in the IMAP Protocol No. ID-BCR: 2007-A00414-49 or IMAP+(n° ID RCB 2011-A01493-38)(see how the study below) have signed forms no objection and consent to study participation

Exclusion Criteria:

Traduction (français > anglais)

* Metastatic
* Cancer of the breast other than primitive
* Patients with paraneoplastic syndrome
* Patients under 45 years
* Patients whose achievement is below level 3 'end of primary schooling "(scale Barbizet)
* Patients with adjuvant chemotherapy is associated with targeted therapy
* Patients who have received other cancer treatments (chemotherapy or radiotherapy brain)
* Contraindication to the implementation of an MRI (claustrophobia, metal objects in the body)
* disorders of higher functions existing in the administration of chemotherapy
* Neurologic earlier
* Pathology psychiatric evolutionary
* Refusal of participation
* Patients unable to meet the cognitive tests
* Drug use
* Heavy drinking

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Assess the relationship between memory impairment and brain dysfunction | Before chemotherapy (baseline), end of chemotherapy and follow-up up to 12 months after chemotherapy
  The main objective is to assess the relationship between memory impairment and brain dysfunction in patients treated with adjuvant chemotherapy for breast cancer (before and after treatment), compared to a group of healthy subjects.

SECONDARY OUTCOMES:
Impact of age | Before chemotherapy (baseline), end of chemotherapy and follow-up up to 12 months after chemotherapy
  The secondary objective is to assess the impact of age on the extent of memory impairment.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre de recherche CYCERON, Caen, Calvados
  - Centre François BACLESSE, Caen, Calvados